CLINICAL TRIAL: NCT03576469
Title: A Single-site, Open-Label, Pilot Study to Evaluate the Benefit of RUCONEST® in Subjects Who Experience ADRs Related to IVIG Infusions
Brief Title: A Study to Evaluate the Benefit of RUCONEST® in Subjects Who Experience ADRs Related to IVIG Infusions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IMMUNOe Research Centers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIS201702-CVID
Record Dates: First submitted 2018-06-15; First posted 2018-07-03 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: CVI - Common Variable Immunodeficiency
Keywords: Intravenous Immunoglobulin; C1-esterase inhibitor; Adverse drug reaction (ADR)
MeSH Terms: conditions — Common Variable Immunodeficiency; Angioedemas, Hereditary; Drug-Related Side Effects and Adverse Reactions | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- C1-esterase inhibitor [recombinant] (C1-INH-R) (Experimental): Single-site, open-label arm to evaluate the benefit of C1-INH-R in subjects on IVIG therapy who experience ADRs. The study will have 2 periods:
  * 6 - 8 weeks - subjects will receive 2 infusions of IVIG
  * 9 - 12 weeks - subjects will receive 3 infusions of C1-INH-R prior to IVIG infusion
  Interventions: Biological: C1-esterase inhibitor [recombinant] (C1-INH-R)

INTERVENTIONS:
Biological: C1-esterase inhibitor [recombinant] (C1-INH-R) — C1-INH-R is FDA approved and indicated for the treatment of acute attacks of angioedema in adolescent and adult patients with Hereditary Angioedema (HAE) as a replacement for low levels of C1-esterase inhibitor or low function of C1-esterase inhibitor

SUMMARY:
Patients receiving intravenous immunoglobulin (IVIG) therapy for primary immunodeficiency and neurologic conditions may experience adverse drug reactions (ADRs). The mechanism of the ADR is unknown. Currently, the standard practice for these patients is to change from IV to subcutaneous IG (SCIG) but because of the need of immunomodulation or patient preference, SCIG may not be an option. Data has shown that some levels of complement decrease from pre- to post-infusion of IVIG. This study is to determine if replacing this complement protein may ameliorate ADRs.

DETAILED DESCRIPTION:
This is a single-site, pilot study conducted in the US to determine the benefit of human C1-esterase inhibitor [recombinant] (C1-INH-R) therapy to ameliorate ADRs in subjects receiving IVIG therapy experience ADRs post-infusion. Subjects who are currently receiving IVIG for immunodeficiency or neurologic conditions and experience ADRs will be enrolled.

In part 1, subjects will continue to receive IVIG for two infusions. Complement proteins will be measured pre- and post-infusion. Quality of life and other questionnaires will be administered.

In part 2, subjects will receive C1-INH-R infusion prior to receiving IVIG infusion for three infusions. Complement proteins will be measured pre- and post- infusion. Quality of life and other questionnaires will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older experiencing ADRs related to IVIG infusions
* Stable dose of IVIG for 3 months
* Willing to comply with all aspects of the protocol, including blood draws
* Female patients of childbearing potential who are sexually active must be willing to use an acceptable form of contraception. Acceptable forms of contraception are defined as those with a failure rate < 1% when properly applied and include: a combination oral pill, some intra-uterine devices, and a sterilized partner in a stable relationship. Female patients must not be pregnant, planning to become pregnant, or be actively breastfeeding through the entire study period.

Exclusion Criteria:

* Receiving treatment for HAE, either prophylactic or acute therapy
* Patients with medical history of allergy to rabbits or rabbit-derived products (including rhC1INH)
* Patients who are pregnant, or breastfeeding, or are currently intending to become pregnant.
* Patients who, in the investigator's opinion, might not be suitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The change in Modified Fatigue Severity Scale (mFSS) | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Subject-rated Rasch-built 7-item modified fatigue survey scale. Scale rated 0 - 3 (3 = agree, 0 = less agree)
The change in Modified Fatigue Impact Scale (MFIS) | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Subject-rated 24 item questionnaire measuring the impact of fatigue rated 0 - 4 (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = almost always)
The change in Migraine Disability Assessment (MIDAS) | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Headache severity measurement of number of days affected after infusion
The change in Headache Impact Scale (HIT-6) | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Subject-rated measurement of the impact headaches have on the ability to function on the job, at school, at home and in social situations. 6 item questionnaire rated from never (6 points each), rarely (8 points each), sometimes (10 points each), very often (11 points each), always (13 points each). The higher number the more the impact.
The change in Activities of Daily Living Sliding Scale | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Subject-rated 10 point scale measuring level of activity with 1 being the worst (least) and 10 being the best (greatest)
The change in Activities of Daily Living Questionnaire | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Calculates the number of days missed from work, school/daycare/activities, housework, and regular exercise
The change in Energy Sliding Scale | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Subject-rated10 point scale measuring energy level with 1 being the worst (Lowest) and 10 being the best (highest)
The change in Infection Questionnaire | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Subject-rated 7 item infection questionnaire measured from 1 to 10 with 1 being the least affected and 10 being the most affected.
The change in Perceived Deficits Questionnaire - cognitive assessment | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Subject-rated 20 item questionnaire measuring memory, attention and concentration rated 0 to 4 (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = almost always) with the lower score being least impact.
The change in 36 item short form survey (SF-36) | Measurement prior to infusion 3 (week 9 - 12) compared to end of study (week 19 - 25)
  Health Survey asks 36 questions to measure functional health and well-being from the patient's point of view.
Change in the number of ADRs | Measured at each infusion (every 3 - 4 weeks)
  Adverse reactions to infusions

SECONDARY OUTCOMES:
Change in levels of C1-INH pre- and post-infusion | Measurement at each infusion (every 3 - 4 weeks)
  Laboratory levels of C1-INH total and functional

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Melamed, MD, Principal Investigator — IMMUNOe Research Centers
Locations (1):
- IMMUNOe Research Centers, Centennial, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Melamed IR, Miranda H, Heffron M, Harper JR. Recombinant Human C1 Esterase Inhibitor for the Management of Adverse Events Related to Intravenous Immunoglobulin Infusion in Patients With Common Variable Immunodeficiency or Polyneuropathy: A Pilot Open-Label Study. Front Immunol. 2021 Mar 2;12:632744. doi: 10.3389/fimmu.2021.632744. eCollection 2021. PMID 33737935